CLINICAL TRIAL: NCT03530007
Title: Comparison Between Two Different Doses of Ondansetron on the Incidence of Spinal Shivering During Cesarean Section
Brief Title: Anti-shivering Effect of Ondansetron
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdel-Baky Abdel-Rahman, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00008718/3167
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Shivering; Ondansetron
MeSH Terms: interventions — Saline Solution; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- normal saline (Active Comparator): patients received normal saline for prevention of shivering during spinal anesthesia
  Interventions: Drug: Normal saline
- ondansetron 4MG (Active Comparator): patients received 4 mg of ondansetron for prevention of spinal shivering
  Interventions: Drug: Ondansetron 4 MG
- ondansetron 8MG (Active Comparator): patients received 8 mg of ondansetron for prevention of spinal shivering
  Interventions: Drug: Ondansetron 8mg

INTERVENTIONS:
Drug: Normal saline — normal saline used for prevention of spinal shivering
  Other Names: placebo
  Arms: normal saline
Drug: Ondansetron 4 MG — ondansetron 4 MG used for prevention of spinal shivering
  Other Names: low ondansetron
  Arms: ondansetron 4MG
Drug: Ondansetron 8mg — ondansetron 8 MG used for prevention of spinal shivering
  Other Names: high ondansetron
  Arms: ondansetron 8MG

SUMMARY:
Shivering is one of the most frequent complications occurring during or after spinal anesthesia with many side effects. The aim of the present study was to compare between two different doses of ondansetron for anti-shivering effect

DETAILED DESCRIPTION:
Shivering is one of the most frequent complications occurring during or after spinal anesthesia, it affects about 40%-60 % of patients under spinal anesthesia. Intra and Post spinal shivering is distressing for the patients and anesthetist. Shivering may aggravate medical conditions in patients with limited cardiac or respiratory functions. It increases tissue oxygen demand many folds which in turn leads to increase the load on respiratory and cardiac systems to cope with increased aerobic metabolism. Shivering interferes with good patient monitoring by causing artifacts of electrocardiography, invasive and non-invasive blood pressure, pulse oximetry, etc... . Postoperatively shivering may cause discomfort to the patient, increases wound pain by stretching incision, increase the incidence of bleeding and infection.

We aim to compare the prophylactic use of two different doses of ondansetron on the incidence of shivering after spinal anesthesia in patients scheduled for lower limb surgery.

The primary outcome was percentage of patients suffering from shivering after spinal anesthesia, secondary outcomes include any side effects related to both doses.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Both sexes
* American Society of Anesthesiologists
* physical status I and II
* scheduled for lower limb surgery under spinal anesthesia

Exclusion Criteria:

* Uncooperative patients
* psychologically unstable patients
* obese patients with BMI >30 preoperative use of ondansetron, or opioids Fever Patients with some clinical conditions like hypo- or hyperthyroidism, Parkinson's disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
incidence of shivering | for 24 hours after spinal anesthesia
  Incidence of shivering among patients in both groups

SECONDARY OUTCOMES:
Axillary temperature | for 24 hours after spinal anesthesia
  patient temperature measured from axillary site
core temperature | for 24 hours after spinal anesthesia
  patient temperature measured from tympanic site
incidence of hypotension | for 24 hours after spinal anesthesia
  Incidence of hypotension between patients in both groups
incidence of nausea and vomiting | for 24 hours after spinal anesthesia
  Incidence of nausea and vomiting among patients in both groups